CLINICAL TRIAL: NCT02073539
Title: The Method of Proper Chest Compression Depth With Conventional and One Accelerometer Feedback Device During CPR in Hospital
Brief Title: The Manikin Study of Chest Compression With One Accelerometer Feedback Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Lee Sang Hyun, Clinical fellow, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2013-12-010-001
Record Dates: First submitted 2014-02-24; First posted 2014-02-27 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Cardiac Arrest
Keywords: Chest compression; One accelerometer; Manikin Study
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- chest compression with 5cm feedback (Experimental): We will feedback by one accelerometer (U-cpr). U-cpr is android based smartphone application.
  Interventions: Device: Stryker ST104-747; Device: Shinchang SB-34p
- chest compression with 6cm feedback (Experimental): We will feedback by one accelerometer(U-cpr). U-cpr is android based smartphone application.
  Interventions: Device: Stryker ST104-747; Device: Shinchang SB-34p
- chest compression with 7cm feedback (Experimental): We will feedback by one accelerometer(U-cpr). U-cpr is android based smartphone application.
  Interventions: Device: Stryker ST104-747; Device: Shinchang SB-34p

INTERVENTIONS:
Device: Stryker ST104-747 — 760 x 2110 mm, 228 kg, Stryker Co., Kalamazoo, Michigan, US
  Other Names: Transport stretcher®
Device: Shinchang SB-34p — , 850 x 2080 mm,Shinchang Co.,Busan,ROK
  Other Names: Transport stretcher®

SUMMARY:
Chest compression (CC) feedback devices are used to perform CC measurements effectively and accurately on patients in hospital beds. However, these devices do not take account of the compression of the mattress, which results in overestimation of CC depth. This study is the validation study to demonstrate that a new method using one accelerometer(U-cpr) is useful to overcome this limitation and thus measure compression depth more accurately when performing cardiopulmonary resuscitation (CPR) on patients.

DETAILED DESCRIPTION:
Data collection The participants will be divided into three groups by random drawings. Each performer in the three-groups will compress the chest of the manikin on the bed with real-time 5cm,6cm and 7cm feed-back by one accelerometer (U-cpr).We will use two beds [Stryker ST104-747(Transport stretcher®, 760 x 2110 mm, 228 kg, Stryker Co., Kalamazoo, Michigan, US) ,Shinchang SB-34p (Transport stretcher® , 850 x 2080 mm,Shinchang Co.,Busan,ROK)]. Each participants will do 6 cycles of chest compression and 1cyle will be 2minutes. Between each cycles, participants will take a rest 5minutes.

ELIGIBILITY:
Inclusion Criteria:

* Postgraduates year 1,2,3,4 and Emergency physicians in emergency department

Exclusion Criteria:

* Wrist or Low back disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Chest compression depth | Within 1day
  Primary out come is measured by Resusci Anne Modular System Skill Reporter manikin (9.89 kg, Laerdal Medical, Orpington, UK)

SECONDARY OUTCOMES:
Chest compression rate | Within 1day
  Secondary out is measured by Resusci Anne Modular System Skill Reporter manikin (9.89 kg, Laerdal Medical, Orpington, UK).

CONTACTS AND LOCATIONS:
Overall Officials: Sang hyun Lee, M.D, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea